CLINICAL TRIAL: NCT00311402
Title: JASAP: Japanese Aggrenox Stroke Prevention vs. Aspirin Programme, Phase III Study to Compare the Preventive Effect of Recurrent Brain Infarction and Safety of Aggrenox (Combination Drug Containing Sustained-release Dipyridamole 200 mg/Acetylsalicylic Acid 25 mg) Twice Daily vs. Acetylsalicylic Acid 81 mg Once Daily
Brief Title: JASAP: Japanese Aggrenox Stroke Prevention vs. Aspirin Programme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Prevention
Other Study IDs: 9.178
Record Dates: First submitted 2006-03-28; First posted 2006-04-06 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Aspirin, Dipyridamole Drug Combination; Aspirin

ARMS (2):
- Aggrenox Capsule (Other)
  Interventions: Drug: Aggrenox capsule
- Acetylsalicylic Acid (ASA) 81 mg Tablet (Other)
  Interventions: Other: Acetylsalicylic Acid (ASA)

INTERVENTIONS:
Drug: Aggrenox capsule — extended-release dipyridamole 200 mg plus ASA 50 mg in a capsule, 2 capsules twice daily
  Arms: Aggrenox Capsule
Other: Acetylsalicylic Acid (ASA) — Acetylsalicylic Acid (ASA) 81 mg, 1 tablet once daily
  Arms: Acetylsalicylic Acid (ASA) 81 mg Tablet

SUMMARY:
Phase III study to compare the preventive effect of recurrent brain infarction and safety of Aggrenox (combination drug containing sustained-release dipyridamole 200 mg/acetylsalicylic acid 25 mg) twice daily vs. acetylsalicylic acid 81 mg once daily

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of cerebral infarction (excluding cardiogenic cerebral embolism) who meet the diagnostic criteria based on the National Institute of Neurological Disorders and Stroke (NINDS) ad hoc committee's classification of cerebrovascular disease III.

1. Patients who have had an onset of cerebral infarction, the time of which is known, between 1 week and 6 months before the time of enrolment (including first and recurrent cerebral infarctions)
2. Patients who are 50 years or older
3. Patients whose neurological signs and symptoms are considered to be stable by the investigator or sub-investigator
4. Patients with a finding corresponding to the responsible focus confirmed by head X-ray computerised tomography (CT) or magnetic resonance imaging (MRI)
5. Patients who have at least two of the following risk factors:

   * diabetes
   * hypertension (systolic blood pressure is 140 mmHg or higher or diastolic blood pressure is 90 mmHg or higher) or under treatment of hypertension
   * smoker (at the time of onset of cerebral infarction)
   * obesity (Body mass index (BMI) is more than 25 kg/m2)
   * previous vascular disease (stroke, acute myocardial infarction or peripheral arterial disease before the onset of cerebral infarction)
   * end-organ damage (retinopathy, left ventricular hypertrophy (LVH) or microalbuminuria)
   * hyperlipidaemia

Exclusion Criteria:

1. Patients with a diagnosis of brain disorders with a bleeding risk such as brain haemorrhage, subarachnoid haemorrhage, cerebral arteriovenous (AV) malformation, cerebral AV aneurysms and brain tumours
2. Patients with complications of cardiac disorders (atrial fibrillation, mitral valve stenosis, severe cardiac valve disorders) that may provide an embolic source for cerebral embolism
3. Patients having had acute coronary syndromes (acute myocardial infarction, unstable angina) within 6 months after enrolment in this study
4. Patient with hypersensitivity to dipyridamole preparations
5. Patients with a history of drug allergy to acetylsalicylic acid (ASA) or aspirin asthma
6. Patients with a history of peptic ulcer
7. Patients having undergone arterial reconstruction after development of cerebral infarction
8. Patients with very severe impairment (4 or 5 on Modified Rankin Scale)
9. Patients with bleeding or bleeding tendencies (haemophilia, haemorrhage urinary tract, vitreous haemorrhage, etc.)
10. Patients with severe hypertension (systolic blood pressure is 180 mmHg or higher or diastolic blood pressure is 110 mmHg or higher)
11. Patients with complications such as serious cardiac, renal and hepatic disorders
12. Patients with a malignant tumour or having had a tumour treatment in the past 5 years
13. Women who are or may be pregnant or lactating women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1295 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (151):
- Japan (151):
  - 9.178.060 Boehringer Ingelheim Investigational Site, Adachi-ku, Tokyo
  - 9.178.017 Boehringer Ingelheim Investigational Site, Adumino, Nagano
  - 9.178.032 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 9.178.074 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 9.178.062 Boehringer Ingelheim Investigational Site, Ako, Hyogo
  - 9.178.064 Boehringer Ingelheim Investigational Site, Aoba-ku, Yokohama, Kanagawa
  - 9.178.097 Boehringer Ingelheim Investigational Site, Aoi-ku, Shizuoka, Shizuoka
  - 9.178.056 Boehringer Ingelheim Investigational Site, Asahi, Chiba
  - 9.178.067 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 9.178.117 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 9.178.166 Boehringer Ingelheim Investigational Site, Atsugi, Kanagawa
  - 9.178.089 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 9.178.054 Boehringer Ingelheim Investigational Site, Chitose, Hokkaido
  - 9.178.133 Boehringer Ingelheim Investigational Site, Chuo-ku, Chiba, Chiba
  - 9.178.030 Boehringer Ingelheim Investigational Site, Chuo-ku, Kobe, Hyogo
  - 9.178.077 Boehringer Ingelheim Investigational Site, Chuo-ku, Sapporo, Hokkaido
  - 9.178.002 Boehringer Ingelheim Investigational Site, Chuo-Ku, Sappro, Hokkaido
  - 9.178.119 Boehringer Ingelheim Investigational Site, Chuo-ku, Sappro, Hokkaido
  - 9.178.161 Boehringer Ingelheim Investigational Site, Daito, Osaka
  - 9.178.112 Boehringer Ingelheim Investigational Site, Fuchu, Tokyo
  - 9.178.098 Boehringer Ingelheim Investigational Site, Fujieda, Shizuoka
  - 9.178.046 Boehringer Ingelheim Investigational Site, Fukaya, Saitama
  - 9.178.145 Boehringer Ingelheim Investigational Site, Fukui, Fukui
  - 9.178.099 Boehringer Ingelheim Investigational Site, Fukuroi, Shizuoka
  - 9.178.165 Boehringer Ingelheim Investigational Site, Funabashi, Chiba
  - 9.178.072 Boehringer Ingelheim Investigational Site, Fushimi-ku, Kyoto, Kyoto
  - 9.178.081 Boehringer Ingelheim Investigational Site, Gifu, Gifu
  - 9.178.024 Boehringer Ingelheim Investigational Site, Habikino, Osaka
  - 9.178.136 Boehringer Ingelheim Investigational Site, Hachioji, Tokyo
  - 9.178.082 Boehringer Ingelheim Investigational Site, Hakodate, Hokkaido
  - 9.178.118 Boehringer Ingelheim Investigational Site, Hakodate, Hokkaido
  - 9.178.052 Boehringer Ingelheim Investigational Site, Hamada, Shimane
  - 9.178.138 Boehringer Ingelheim Investigational Site, Hashima-gun, Gifu
  - 9.178.169 Boehringer Ingelheim Investigational Site, Hidaka, Saitama
  - 9.178.001 Boehringer Ingelheim Investigational Site, Higashi-ku, Sappro, Hokkaido
  - 9.178.026 Boehringer Ingelheim Investigational Site, Higashi-osaka, Osaka
  - 9.178.163 Boehringer Ingelheim Investigational Site, Higashidakawa-gun, Yamagata
  - 9.178.120 Boehringer Ingelheim Investigational Site, Higashimatsushima, Miyagi
  - 9.178.028 Boehringer Ingelheim Investigational Site, Higashinari-ku, Osaka, Osaka
  - 9.178.140 Boehringer Ingelheim Investigational Site, Higashiosaka, Osaka
  - 9.178.122 Boehringer Ingelheim Investigational Site, Higashisonogi-gun, Nagasaki
  - 9.178.101 Boehringer Ingelheim Investigational Site, Higashiyodogawa-ku, Osaka, Osaka
  - 9.178.093 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 9.178.153 Boehringer Ingelheim Investigational Site, Hitachi, Ibaraki
  - 9.178.005 Boehringer Ingelheim Investigational Site, Hitachinaka, Ibaraki
  - 9.178.079 Boehringer Ingelheim Investigational Site, Ibusuki, Kagoshima
  - 9.178.143 Boehringer Ingelheim Investigational Site, Ichikawa, Chiba
  - 9.178.019 Boehringer Ingelheim Investigational Site, Iida, Nagano
  - 9.178.129 Boehringer Ingelheim Investigational Site, Inashiki-gun, Ibaraki
  - 9.178.011 Boehringer Ingelheim Investigational Site, Isesaki, Gunma
  - 9.178.045 Boehringer Ingelheim Investigational Site, Isesaki, Gunma
  - 9.178.031 Boehringer Ingelheim Investigational Site, Itami, Hyogo
  - 9.178.135 Boehringer Ingelheim Investigational Site, Iwanuma, Miyagi
  - 9.178.104 Boehringer Ingelheim Investigational Site, Iwata, Shizuoka
  - 9.178.095 Boehringer Ingelheim Investigational Site, Izuka, Fukuoka
  - 9.178.080 Boehringer Ingelheim Investigational Site, Izumisano, Osaka
  - 9.178.139 Boehringer Ingelheim Investigational Site, Izumo, Shimane
  - 9.178.113 Boehringer Ingelheim Investigational Site, Izunokuni, Shizuoka
  - 9.178.115 Boehringer Ingelheim Investigational Site, Kahoku-gun, Ishikawa
  - 9.178.147 Boehringer Ingelheim Investigational Site, Kameda-gun, Hokkaido
  - 9.178.092 Boehringer Ingelheim Investigational Site, Kamigyo-ku, Kyoto, Kyoto
  - 9.178.008 Boehringer Ingelheim Investigational Site, Kasama, Ibaraki
  - 9.178.035 Boehringer Ingelheim Investigational Site, Kasuga, Fukuoka
  - 9.178.037 Boehringer Ingelheim Investigational Site, Kasuga, Fukuoka
  - 9.178.051 Boehringer Ingelheim Investigational Site, Kawachinagano, Osaka
  - 9.178.086 Boehringer Ingelheim Investigational Site, Kisarazu, Chiba
  - 9.178.162 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 9.178.102 Boehringer Ingelheim Investigational Site, Kita-ku, Nagoya, Aichi
  - 9.178.023 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka, Osaka
  - 9.178.127 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka, Osaka
  - 9.178.004 Boehringer Ingelheim Investigational Site, Kita-ku, Sappro, Hokkaido
  - 9.178.154 Boehringer Ingelheim Investigational Site, Kitami, Hokkaido
  - 9.178.155 Boehringer Ingelheim Investigational Site, Kitami, Hokkaido
  - 9.178.069 Boehringer Ingelheim Investigational Site, Kiyose, Tokyo
  - 9.178.070 Boehringer Ingelheim Investigational Site, Kiyose, Tokyo
  - 9.178.121 Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - 9.178.141 Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - 9.178.061 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 9.178.085 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 9.178.075 Boehringer Ingelheim Investigational Site, Koshi, Kumamoto
  - 9.178.107 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 9.178.063 Boehringer Ingelheim Investigational Site, Kushiro
  - 9.178.083 Boehringer Ingelheim Investigational Site, Kushiro
  - 9.178.126 Boehringer Ingelheim Investigational Site, Kushiro
  - 9.178.150 Boehringer Ingelheim Investigational Site, Marugame, Kagawa
  - 9.178.164 Boehringer Ingelheim Investigational Site, Matsudo, Chiba
  - 9.178.015 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 9.178.130 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 9.178.057 Boehringer Ingelheim Investigational Site, Meito-ku, Nagoya, Aichi
  - 9.178.013 Boehringer Ingelheim Investigational Site, Midori-ku, Yokohama, Kanagawa
  - 9.178.043 Boehringer Ingelheim Investigational Site, Minami-ku, Hiroshima, Hiroshima
  - 9.178.068 Boehringer Ingelheim Investigational Site, Miyagino-ku, Sendai, Miyagi
  - 9.178.116 Boehringer Ingelheim Investigational Site, Miyazaki, Miyazaki
  - 9.178.142 Boehringer Ingelheim Investigational Site, Moriguchi, Osaka
  - 9.178.078 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 9.178.084 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 9.178.009 Boehringer Ingelheim Investigational Site, Moriya, Ibaraki
  - 9.178.149 Boehringer Ingelheim Investigational Site, Moriya, Ibaraki
  - 9.178.071 Boehringer Ingelheim Investigational Site, Musashimurayama, Tokyo
  - 9.178.012 Boehringer Ingelheim Investigational Site, Musashino, Tokyo
  - 9.178.100 Boehringer Ingelheim Investigational Site, Naka-ku, Hamamatsu, Shizuoka
  - 9.178.110 Boehringer Ingelheim Investigational Site, Naka-ku, Hamamatsu, Shizuoka
  - 9.178.020 Boehringer Ingelheim Investigational Site, Naka-ku, Nagoya, Aichi
  - 9.178.053 Boehringer Ingelheim Investigational Site, Nakagawa-ku, Nagoya, Aichi
  - 9.178.132 Boehringer Ingelheim Investigational Site, Nakagawa-ku, Nagoya, Nagoya
  - 9.178.124 Boehringer Ingelheim Investigational Site, Namegata, Ibaraki
  - 9.178.158 Boehringer Ingelheim Investigational Site, Nanao, Ishikawa
  - 9.178.029 Boehringer Ingelheim Investigational Site, Nishi-yodogawa-ku, Osaka, Osaka
  - 9.178.096 Boehringer Ingelheim Investigational Site, Nishisonogi-gun, Nagasaki
  - 9.178.087 Boehringer Ingelheim Investigational Site, Noda, Chiba
  - 9.178.058 Boehringer Ingelheim Investigational Site, Obu, Aichi
  - 9.178.034 Boehringer Ingelheim Investigational Site, Ohnojo, Fukuoka
  - 9.178.157 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 9.178.167 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 9.178.137 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 9.178.027 Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - 9.178.073 Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - 9.178.018 Boehringer Ingelheim Investigational Site, Saku, Nagano
  - 9.178.160 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 9.178.041 Boehringer Ingelheim Investigational Site, Setagaya-ku, Tokyo
  - 9.178.088 Boehringer Ingelheim Investigational Site, Shibuya-ku, Tokyo
  - 9.178.022 Boehringer Ingelheim Investigational Site, Shimogyo-ku, Kyoto, Kyoto
  - 9.178.076 Boehringer Ingelheim Investigational Site, Shimotsuke, Tochigi
  - 9.178.055 Boehringer Ingelheim Investigational Site, Shiroishi, Miyagi
  - 9.178.111 Boehringer Ingelheim Investigational Site, Simizu-ku, Shizuoka, Shizuoka
  - 9.178.151 Boehringer Ingelheim Investigational Site, Suminoe-ku, Osaka, Osaka
  - 9.178.156 Boehringer Ingelheim Investigational Site, Susono, Shizuoka
  - 9.178.014 Boehringer Ingelheim Investigational Site, Suwa, Nagano
  - 9.178.039 Boehringer Ingelheim Investigational Site, Takasaki, Gunma
  - 9.178.146 Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - 9.178.144 Boehringer Ingelheim Investigational Site, Takayama, Gifu
  - 9.178.003 Boehringer Ingelheim Investigational Site, Takikawa, Hokkaido
  - 9.178.040 Boehringer Ingelheim Investigational Site, Tatebayashi, Gunma
  - 9.178.066 Boehringer Ingelheim Investigational Site, Teine-ku, Sapporo, Hokkaido
  - 9.178.134 Boehringer Ingelheim Investigational Site, Tenri, Nara
  - 9.178.159 Boehringer Ingelheim Investigational Site, Tonami, Toyama
  - 9.178.007 Boehringer Ingelheim Investigational Site, Toride, Ibaraki
  - 9.178.047 Boehringer Ingelheim Investigational Site, Toyama, Toyama
  - 9.178.090 Boehringer Ingelheim Investigational Site, Toyohashi, Aichi
  - 9.178.131 Boehringer Ingelheim Investigational Site, Toyota, Aichi
  - 9.178.006 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki
  - 9.178.016 Boehringer Ingelheim Investigational Site, Ueda, Nagano
  - 9.178.091 Boehringer Ingelheim Investigational Site, Uji, Kyoto
  - 9.178.050 Boehringer Ingelheim Investigational Site, Ukyo-ku, Kyoto, Kyoto
  - 9.178.106 Boehringer Ingelheim Investigational Site, Urayasu, Chiba
  - 9.178.148 Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
  - 9.178.114 Boehringer Ingelheim Investigational Site, Wko, Saitama
  - 9.178.152 Boehringer Ingelheim Investigational Site, Yaizu, Shizuoka
  - 9.178.125 Boehringer Ingelheim Investigational Site, Yamashina, Kyoto, Kyoto
  - 9.178.108 Boehringer Ingelheim Investigational Site, Yanai, Yamaguchi
  - 9.178.103 Boehringer Ingelheim Investigational Site, Yao, Osaka

REFERENCES:
- [Derived] Uchiyama S, Ikeda Y, Urano Y, Horie Y, Yamaguchi T. The Japanese aggrenox (extended-release dipyridamole plus aspirin) stroke prevention versus aspirin programme (JASAP) study: a randomized, double-blind, controlled trial. Cerebrovasc Dis. 2011;31(6):601-13. doi: 10.1159/000327035. Epub 2011 Apr 19. PMID 21502757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment initiated from June 2006 and completed in December 2007.
Groups:
- Aggrenox Capsule: Aggrenox (extended-release dipyridamole 200 mg plus ASA 50 mg in a capsule), 2 capsules twice daily
- Acetylsalicylic Acid (ASA) 81 mg Tablet: ASA 81 mg, 1 tablet once daily
Period: Overall Study
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Started | 655 | 639
Completed | 445 | 462
Not Completed | 210 | 177
Not completed — Adverse Event | 118 | 105
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 17 | 18
Not completed — Lack of Efficacy | 58 | 42
Not completed — Protocol Violation | 7 | 6
Not completed — IRB's rejection etc. | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet | Total
Number analyzed (Participants) | 655 | 639 | 1294
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.1) | 66.0 (8.6) | 66.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 186 | 369
  Male | 472 | 453 | 925

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With First Recurrent Cerebral Infarction (Fatal or Non-fatal)
Description: All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: All outcomes and efficacy endpoints were analysed on the basis of the full analysis set (FAS). FAS population excluded that 1) patients who did not meet inclusion criteria, 2) patients who had never taken the investigational products, and 3) patients who had no data after drug administration.
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 45 | 32
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; Non-event rate was calculated by using the Kaplan-Meier method and the comparison of groups was made by using the Cox proportional hazard regression model; Test type: Non-Inferiority or Equivalence — The non-event rates after 1 year in the Aggrenox group and ASA group are estimated at 94.0% and 91.5%, respectively. The non-inferiority margin was set to 2%. Under these conditions, 500 patients per group were supposed to be enough to detect the non-inferiority of Aggrenox with over 80% power; p = 0.097, Regression, Cox; Cox Proportional Hazard = 1.47, 95% CI [0.93 to 2.31]

2. Secondary Outcome: Number of Patients With Brain (Cerebral) Haemorrhage
Description: All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 12 | 7
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.223, Regression, Cox; Cox Proportional Hazard = 1.79, 95% CI [0.70 to 4.54]

3. Secondary Outcome: Number of Patients With Subarachnoid Haemorrhage
Description: All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 0 | 1
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.998, Regression, Cox; Cox Proportional Hazard = 0, 95% CI 1-sided [lower limit 0]

4. Secondary Outcome: Number of Patients With Transient Ischemic Attack (TIA)
Description: All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 3 | 3
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.977, Regression, Cox; Cox Proportional Hazard = 1.02, 95% CI [0.21 to 5.07]

5. Secondary Outcome: Number of Patients With Acute Coronary Syndrome (ACS)
Description: ACS contains acute myocardial infarction (MI), unstable angina and sudden cardiac death. All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 9 | 16
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.192, Regression, Cox; Cox Proportional Hazard = 0.58, 95% CI [0.26 to 1.31]

6. Secondary Outcome: Number of Patients With Other Vascular Events
Description: This endpoints were defined as pulmonary embolism, retinal vascular disorder, deep vein thrombosis, peripheral artery obstruction and vascular intervention. All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 11 | 6
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.215, Regression, Cox; Cox Proportional Hazard = 1.88, 95% CI [0.69 to 5.07]

7. Secondary Outcome: Number of Patients With Ischemic Vascular Event Composite Endpoint
Description: This is a composite endpoint of cerebral infarction, transient ischemic attack (TIA), acute myocardial infarction (MI), unstable angina and sudden death attributable to thromboembolism. All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 57 | 51
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.443, Regression, Cox; Cox Proportional Hazard = 1.16, 95% CI [0.79 to 1.69]

8. Post Hoc Outcome: Number of Patients With Stroke
Description: This is a composite endpoint of cerebral infarction, brain (cerebral) hemorrhage and subarachnoid haemorrhage. All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 57 | 39
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.043, Regression, Cox; Cox Proportional Hazard = 1.52, 95% CI [1.01 to 2.29]

9. Post Hoc Outcome: Number of Patients With Intracranial Haemorrhage
Description: All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 13 | 13
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.919, Regression, Cox; Cox Proportional Hazard = 1.04, 95% CI [0.48 to 2.25]

10. Post Hoc Outcome: Number of Patients With Composite Endpoint of Stroke or Major Bleeding
Description: This is a composite endpoint of cerebral infarction, brain (cerebral) hemorrhage, subarachnoid haemorrhage and major bleeding. All events reported by investigators were adjudicated by the independent event assessment committee in a blinded manner.
Time Frame: Up to 124 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Number analyzed (Participants) | 652 | 639
patients | 71 | 55
Statistical Analysis 1: Comparison: Aggrenox Capsule vs Acetylsalicylic Acid (ASA) 81 mg Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.101, Regression, Cox; Cox Proportional Hazard = 1.34, 95% CI [0.94 to 1.91]

ADVERSE EVENTS:
Time Frame: From day of first drug dose until 6 days after last dose, up to 874 days
Arm/Group | Aggrenox Capsule | Acetylsalicylic Acid (ASA) 81 mg Tablet
Serious Adverse Events (participants affected / at risk) | 178/655 | 167/639
Other Adverse Events (participants affected / at risk) | 634/655 | 604/639
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aggrenox Capsule (N=655) | Acetylsalicylic Acid (ASA) 81 mg Tablet (N=639)
Pneumonia (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pleurisy viral (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hyperadrenalism (Endocrine disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 46 | 32
Cerebral haemorrhage (Nervous system disorders) | 5 | 2
Cerebellar haemorrhage (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 3
Thalamus haemorrhage (Nervous system disorders) | 2 | 3
Epilepsy (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Basilar migraine (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1
Putamen haemorrhage (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 6
Maculopathy (Eye disorders) | 0 | 2
Eyelid ptosis (Eye disorders) | 1 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 2
Auricular perichondritis (Ear and labyrinth disorders) | 0 | 1
Vertigo labyrinthine (Ear and labyrinth disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 6
Angina pectoris (Cardiac disorders) | 5 | 4
Myocardial infarction (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 11 | 8
Inguinal hernia (Gastrointestinal disorders) | 1 | 4
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Sudden death (General disorders) | 1 | 4
Multi-organ failure (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Implant site inflammation (General disorders) | 1 | 0
Mass (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema due to renal disease (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 4
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 3
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Blast injury (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Diffuse axonal injury (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aggrenox Capsule (N=655) | Acetylsalicylic Acid (ASA) 81 mg Tablet (N=639)
Nasopharyngitis (Infections and infestations) | 281 | 261
Headache (Nervous system disorders) | 293 | 187
Dizziness (Nervous system disorders) | 58 | 55
Hypertension (Vascular disorders) | 37 | 53
Diarrhoea (Gastrointestinal disorders) | 78 | 42
Constipation (Gastrointestinal disorders) | 34 | 60
Nausea (Gastrointestinal disorders) | 40 | 42
Eczema (Skin and subcutaneous tissue disorders) | 30 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 58 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 39
Fall (Injury, poisoning and procedural complications) | 58 | 69
Contusion (Injury, poisoning and procedural complications) | 46 | 60
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 46 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract